CLINICAL TRIAL: NCT04460534
Title: Detection of SARS-CoV-2 in the Semen of COVID+ Patients (Positive RT-PCR on a Nasopharyngeal Swab)
Brief Title: Detection of COVID-19 (SARS-CoV-2) in the Semen of COVID+ Patients (Positive RT-PCR on a Nasopharyngeal Swab)
Acronym: COVISPERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A01206-33
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: COVID
MeSH Terms: interventions — Diagnosis

STUDY DESIGN:
Intervention Model Description: This is a prospective monocentric, open-label, prospective study of male patients with CoV-2-SARS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COHORT (Experimental): Cohort
  Interventions: Diagnostic Test: diagnostic

INTERVENTIONS:
Diagnostic Test: diagnostic — The principle of this study is to propose to patients in whom a COVID-19 infection is suspected and who are screened for the disease, the joint search for the virus in the semen.

SUMMARY:
The objective of this study is to look for the presence of SARS-CoV-2 in the semen of patients diagnosed with COVID+ based on RT-PCR analysis of nasopharyngeal swabs.

DETAILED DESCRIPTION:
This is a prospective monocentric, open-label, prospective study of male patients with CoV-2-SARS.

ELIGIBILITY:
Inclusion Criteria:

* Male patient between the ages of 18 and 65 who has read and signed the consent form for participation in the study.
* Outpatient or inpatient without signs of respiratory severity, likely to be mobile
* Patient whose medical condition warrants screening for COVID-19 by nasopharyngeal swab

Exclusion Criteria:

* Patient under protective custody, guardianship or trusteeship
* Patient not affiliated to the French social security system
* Inability to provide the subject with informed information and/or written informed consent: dementia, psychosis, consciousness disorders, non-French speaking patient

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Semen collection
Enrollment: 52 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Testing for the presence of COVID-19 (SARS-CoV-2 virus) in the semen | 48 hours
  The search for the SARS-CoV-2 virus in semen will be carried out by RT-PCR analysis with the RealStar kit developed by Altona Diagnostics. The extraction of the nucleic acid suitable for sperm uses the Pure MagNA technique (Diagnostics ROCHE). This is an extraction technique that has already been validated for HIV-type RNA viruses in semen.
  The biological samples will be analysed either during the study or bio-banked and analysed at the end of the study. Only semen samples from patients detected positive for SARS-CoV-2 by RT-PCR on nasopharyngeal swab will be analyzed.
Kinetics of SARS-CoV-2 virus presence in the semen | 1 month
  Patients who have been found to carry the SARS-CoV-2 virus in their semen will be recalled after one month to re-test for the virus. In case of a positive re-test, a new search will be scheduled and so on until a negative result is found.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie DELAROCHE, Pharm D, Principal Investigator — Hôpital privé de Parly II
Locations (1):
- Hôpital Privé de Parly II, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No